CLINICAL TRIAL: NCT00257569
Title: Evaluation of the Efficacy and Safety of Cetirizine Dry Syrup in Children -Suffering From Atopic Dermatitis-
Brief Title: Study Of Atopic Dermatitis In Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104913
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic; Pediatric; Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetirizine Dry Syrup

SUMMARY:
To verify of cetirizine dry syrup to ketotifen dry syrup in the change in the severity of pruritus of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as atopic dermatitis
* Giving informed consent
* Children who have 2 grades or more pruritus score.
* Children who require the treatment with external steroid preparation other than face and head.
* Children with a pruritus severity of 2.
* Mild or severe on the fist day of the treatment period.

Exclusion criteria:

* have spastic disease such as epilepsy
* have a history of drug hypersensitivity
* are lactating or possibly pregnant female Children
* have a skin infection, or with zooparasite such as scabies and pediculosis
* cannot avoid the use of external steroid classified into strong, strongest or very strong
* have eczematous otitis externa with perforation in the eardrum
* have dermal ulcer, or profound heat burn or frostbite of the severity higher than the grade 2
* have asthma that requires the treatment with corticosteroid
* have pruritus only on face and head
* have inappropriate complication of dermal disorder that may influence on the evaluation of the study drug
* are undergoing specific desensitization therapy or immunomodulation therapy or phototherapy.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278
Dates: Start 2005-08

PRIMARY OUTCOMES:
change in the severity of pruritus

SECONDARY OUTCOMES:
-changes in the total pruritus score -daily main pruritus score -improvement of area with pruritus -patient global improvement -Cetirizine serum concentrations -Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site